CLINICAL TRIAL: NCT04637113
Title: Singapore's Health Outcomes After Critical Illness in Kids: the SHACK Study: A Longitudinal Mixed-methods Study in Singapore to Explore the Health Outcomes of Children and Their Parents in the First Six Months After PICU Discharge
Brief Title: Singapore's Health Outcomes After Critical Illness in Kids
Acronym: SHACK
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: University of Plymouth (Other)
Responsible Party: Sponsor
Other Study IDs: theSHACKStudy:Singapore
Record Dates: First submitted 2020-10-14; First posted 2020-11-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Pediatric ALL; Critical Illness; Post Intensive Care Unit Syndrome
Keywords: critical illness; family; race; ethnicity; health outcomes
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients admitted to the PICU meeting eligible criteria: This is a non-interventional study.
  Interventions: Other: This is a non-interventional study

INTERVENTIONS:
Other: This is a non-interventional study — This is a non-interventional study.

SUMMARY:
What is the problem? Every year about 2.5 million children are affected by critical illness and require admission to the pediatric intensive care unit (PICU). However, both children and their parents may encounter difficulties after critical illness. Children affected physically may have difficulties in breathing, eating, and drinking. Parents have reported feeling symptoms of stress such as nightmares and excessive worries after PICU discharge. Currently, the investigators do not know when and how the problems unfold and what harm does it cause. Without this information, healthcare professionals are not equipped to support these families after PICU discharge.

Research Plan? To understand how critical illness could affect the physical, emotional, and social experiences of children age 1 month to 18 years of age and their parents in the first 6 months after a PICU admission.

144 children and their parents will be followed from the time of PICU admission to 6 months after discharge. Children and their parents will complete surveys to measure physical, social, emotional and function outcomes. A total of 12 families will be interviewed at 1 and 3 months after PICU discharge. Using the data provided to map out any trend or changes in this information over time.

Why is this study important? To better understand the experience and health consequences of children and their parents in the first six months after PICU admission. This information would help to identify potential areas to improve the negative consequence of children and their families after a severe illness. Results will be shared to the PICU survivors and their families, national organizations, international pediatric intensive care community to improve the experiences and health outcomes following a PICU admission.

ELIGIBILITY:
Child inclusion criteria:

* Aged 1 month to 18 years at the point of PICU admission
* PICU total length of stay (LOS) ≥ 48 hours at the point of PICU discharge

Parents inclusion criteria:

* (a) Parent or legal guardian; (b) cohabits with the child
* For the family home to be the planned location following hospital discharge.

Exclusion Criteria:

* Opted for a "Do Not Resuscitate" status for their child and/or
* Had participated in the current study in a previous PICU admission within the recruitment period.

Ages: 1 Month to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children age 1 month to 18 years old requiring PICU admission for ≥ 48 hours and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
To describe and compare the change in total score of the Paediatric Quality of Life Inventory Version 4.0 (PedsQL™) in children at baseline from 6 months after PICU discharge. | baseline and 6 months
  The PedsQL instrument consists of 23 items that evaluate 4 domains: physical, emotional, social, and school functioning with summary scores available for physical and psychological health. It is scored using a 5-point Likert scale from 0 (never) to 4 (A lot) with a possible score of 0 to 100.

SECONDARY OUTCOMES:
To determine the correlation between race/ethnicity, children's health baseline, and PICU factors with a total score of the Paediatric Quality of Life Inventory Version 4.0 (PedsQL™) after PICU discharge. | 6 months
  The Paediatric Quality of Life Inventory Version 4.0 (PedsQL™) total score will be used to compare the difference between Chinese, Malay, and Indian families. This instrument consists of 23 items that evaluate 4 domains: physical, emotional, social, and school functioning with summary scores available for physical and psychological health. It is scored using a 5-point Likert scale from 0 (never) to 4 (A lot) with a possible score of 0 to 100.
To investigate the risk factors for parental PTSD using the PTSD Checklist for DSM-5 (PCL-5) six months after their child's' PICU discharge. | 6 months
  PTSD Checklist for DSM-5 (PCL-5) assesses the 20 Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition (DSM-5) symptoms of post-traumatic stress disorder. The 20 items self-report measure is scored on a rating a 5-point Likert scale from 0 (Not at all) to 4 (Extremely). The symptoms severity score ranges from 0-80. A cut-off score between 31-33 is indicative of probable PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fen Poh, Principal Investigator — KK Women's and Children's Hospital, Singapore
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manning JC, Pinto NP, Rennick JE, Colville G, Curley MAQ. Conceptualizing Post Intensive Care Syndrome in Children-The PICS-p Framework. Pediatr Crit Care Med. 2018 Apr;19(4):298-300. doi: 10.1097/PCC.0000000000001476. PMID 29406379
- [Result] Abela KM, Wardell D, Rozmus C, LoBiondo-Wood G. Impact of Pediatric Critical Illness and Injury on Families: An Updated Systematic Review. J Pediatr Nurs. 2020 Mar-Apr;51:21-31. doi: 10.1016/j.pedn.2019.10.013. Epub 2019 Dec 23. PMID 31874458
- [Derived] Poh PF, Lee JH, Sultana R, Manning JC, Carey MC, Latour JM. Physical, Cognitive, Emotional, and Social Health Outcomes of Children in the First 6 Months After Childhood Critical Illness: A Prospective Single-Center Study. Pediatr Crit Care Med. 2024 Dec 1;25(12):1138-1149. doi: 10.1097/PCC.0000000000003622. Epub 2024 Oct 11. PMID 39630545
- [Derived] Poh PF, Lee JH, Manning JC, Carey MC, Sultana R, Latour JM. Singapore's health outcomes after critical illness in kids: A study protocol exploring health outcomes of families 6 months after critical illness. J Adv Nurs. 2021 Aug;77(8):3531-3541. doi: 10.1111/jan.14911. Epub 2021 Jun 3. PMID 34081353